CLINICAL TRIAL: NCT03128385
Title: Comparative Efficacy Research of Intensive and Distributed Constraint-Induced Therapy: Evidence-Based Neurorehabilitation in Children With CP
Brief Title: Evidence-Based Neurorehabilitation in Children With CP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201701011RINC
Record Dates: First submitted 2017-04-18; First posted 2017-04-25 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Cerebral Palsy
Keywords: Upper limb neurorehabilitation; Neurological rehabilitation; Upper extremity
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive CIT Model Program (Experimental): In day camp model, the therapist will monitor and modify the activities to fit each child's ability and need (e.g. implementing task analysis, grading the challenge for each individual with varying capabilities) to make sure the intervention quality is equivalence to the individualized treatment.The day camp model will be arranged as "Adventure Camp" that decorating the treatment place as the adventure world and the participants take role as a warrior. This novel design is mean to enhance and motivate the engagement of participation.
  Interventions: Other: Intensive CIT Model Program
- Distributed CIT Model Program (Experimental): All treatment activities will be focused on the training of the more affected upper limbs with contextual restraint. Investigators choose this child-friendly way to restraint children's non or less impaired hand without any devices. Investigators will provide a unilateral activities and verbal cues to restraint participants' non or less affected side. All tailored activities will be designed as fun and age-appropriated based on the child's preference and parents' concerns. In order to help children to generalize the therapeutic gains to the real world environment, the intervention will take place in the natural environment such as home or school where it may be easier to identify real practical problems and makes the family or caregivers involved more closely and directly.
  Interventions: Other: Distributed CIT Model Program

INTERVENTIONS:
Other: Intensive CIT Model Program — Day Camp Model:
  1. The treatment was delivered in group-based design, 6 hours a day for 6 days (36 hours in total)
  2. constraint of the unaffected hand to encourage the use of the affected hand
  3. massed and repetitive practice of the affected hand during the period of constraint
  4. use of behavioral techniques termed "shaping" to train the affected hand
  Arms: Intensive CIT Model Program
Other: Distributed CIT Model Program — Home-Based Model:
  1. The participants will receive individualized interventions, 2.25 hours a day, two times a week for 8 weeks (36 hours in total).
  2. constraint of the unaffected hand to encourage the use of the affected hand
  3. massed and repetitive practice of the affected hand during the period of constraint
  4. use of behavioral techniques termed "shaping" to train the affected hand
  Arms: Distributed CIT Model Program

SUMMARY:
This 3-year research project aims to investigate and compare the treatment effectiveness (in terms of motor and psychosocial outcomes) and potential predictors (in terms of demographical, biological and psychosocial domains) of the intensive and distributed Child- and Family-Friendly CIT protocols with an equivalent intervention period in children with CP by quasi randomized controlled study design. In addition, the selection and examination of outcome measures were based on the ICF-CY model to provide comprehensively documents.

DETAILED DESCRIPTION:
Upper limb dysfunction is a common and disabling consequence of children with cerebral palsy (CP). As children with hemiplegia primarily have one better funcitoning side of their body and one more affected side, they often tend not to use the affected extremity resulting in the phenoema of developmental disregard. Recent evidence suggests that constraint-induced therapy (CIT) is the most effective technique to improve the use of the affected hand and reduce the developmental disregard in children with CP. However, despite the cumulative evidence supporting the effects of pediatric CIT, the concerns of feasibility and gaps of current knowledge prompt us to conduct this current proposal. The concerns of the feasibility include this approach is emotionally problematic at early stages and researchers suggested that the orginal CIT protocols may be too intrusive for children and their families. The gaps of current knowledge include: no study has directly investigated the effectiveness differences between various CIT models; no study examines, monitors and compares the psychosocial outcomes while receiving the CIT protocols for children and their parents systematically and comprehensively; and no study investigates the possible clinical characteristics of children that may influence the training effects of the various CIT models.

Investigators will recruit a total of 60 children with CP from the CP Association, medical centers, and special educational systems and participants will be assigned to the two intervention groups. The intensive CIT is delivered by the group-based design with 6 hours a day for 6 days (36 hours in total) and the distributed CIT will be delivered by individualized home-based intervention with 2.25 hours a day, two times a week, for 8 weeks (36 hours in total).

ELIGIBILITY:
The inclusion criteria of this study are:

1. aged between 5 and 13 years
2. diagnosed with congenital hemiplegic or children with CP with one more affected side
3. apparently disuse phenomenon of the more affected hand at spontaneous contexts

Participants will be exclude for:

1. excessive muscle tone (Modified Ashworth Scale ≤ 2 at any joints of the upper limb) before beginning treatment
2. severe cognitive, visual, or auditory disorders according to medical documents, parental reports, and the examiner's clinical observation
3. injections of botulinum toxin type A or operations on the UE within 6 months

Ages: 5 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
"change" Melbourne Assessment 2 (MA2) | Intensive and CIT Model Program: baseline, 1 week, 2 months, 6 months; Distributed CIT Model Program: baseline, 1 months, 2 months, 6 months
  The MA2 was developed to investigate the objective upper-limb movement in children with CP aged 2.5 to 15 years (Randall, Imms, Carey, & Pallant, 2014). The test comprises 14 functional tasks (e.g., grasping a pellet, pointing, and etc), which are representative of the most important components of unilateral upper limb function, including reach, grasp, release, and manipulate.
"change" Box and Block Test (BBT) | Intensive and CIT Model Program: baseline, 1 week, 2 months, 6 months; Distributed CIT Model Program: baseline, 1 months, 2 months, 6 months
  The BBT assesses manual dexterity by county the number of blocks that are transferred with a single hand from one compartment to another within 60 seconds. In recent years, it has increasingly been used to assess gross manual dexterity of the affected versus the non-affected hand in children and young adolescents with hemiplegia cerebral palsy.
"change" Pediatric Motor Activity Log-Revised (PMAL-R) | Intensive and CIT Model Program: baseline, 1 week, 2 months, 6 months; Distributed CIT Model Program: baseline, 1 months, 2 months, 6 months
  The PMAL-R is adapted from the Pediatric Motor Activity Log (Taub et al., 2004), which was developed as an outcome measure for evaluating the effectiveness of CIT in children with CP. It is a parent-reported evaluative tool used to capture the spontaneous use of the affected upper limb in 22 daily activities. Each activity is rated by parents/careers on two set (how often and how well) of 6-point ordinal scales (0-5). The 'how often' scale measures amount of use, and the 'how well' scale measures quality of movement, of the affected upper limb. The PMAL-R testing manual is available online.

SECONDARY OUTCOMES:
"change" Bruininks-Oseretsky Test of Motor Proficiency, Second Edition (BOT-2) | Intensive and CIT Model Program: baseline, 1 week, 2 months, 6 months; Distributed CIT Model Program: baseline, 1 months, 2 months, 6 months
  The BOT-2 is widely used as an efficient and standardized measurement of motor control skills for children aged 4 through 21. The subtest 3 of the BOT-2, manual dexterity (MD), will be used to assess a child's upper limb dexterity. The subtests 3 of the BOT-2 consist of 5 goal-directed activities that involve reaching, grasping, and bimanual coordination with small objects to investigate a child's upper limb manual function
"change" Motion Analysis | Intensive and CIT Model Program: baseline, 1 week, 2 months, 6 months; Distributed CIT Model Program: baseline, 1 months, 2 months, 6 months
  For the performance outcome measures, endpoint variables during reach-to-grasp task, namely reaction time, movement time, movement unit, peak velocity and its time percentage during the movement time will be calculated using the wrist marker. For the performance production measures, joint angles of the shoulder, elbow and wrist during reach-to-grasp task will also be calculated to represent the motor strategy of children with CP before and after intervention.
"change" ABILHAND-Kids | Intensive and CIT Model Program: baseline, 1 week, 2 months, 6 months; Distributed CIT Model Program: baseline, 1 months, 2 months, 6 months
  The ABILHAND-Kids questionnaire is a Rasch-based assessment that measures children's perceived difficulty in performing ADL that require the use of the bilateral upper limbs. It contains 21 items measuring manual ability and is rated on a 3-point response scale. The parent is asked to fill in the questionnaire by estimating their child's ease or difficulty in performing each activity, irrespective of the limb(s) the child actually use and whatever the strategies used to perform the activity.
"change" Pediatric Evaluation of Disability Inventory (PEDI) | Intensive and CIT Model Program: baseline, 1 week, 2 months, 6 months; Distributed CIT Model Program: baseline, 1 months, 2 months, 6 months
  The PEDI is used to evaluate the generalization of treatment effect to daily life. The PEDI assesses the level of independence in daily activities in children with cerebral palsy, including the functional performance and level of assistance needed in daily activities.
"change" Dimensions of Mastery Questionnaire (DMQ) | Intensive and CIT Model Program: baseline, 1 week, 2 months, 6 months; Distributed CIT Model Program: baseline, 1 months, 2 months, 6 months
  The DMQ provides a primary caregiver's perceptions of mastery motivation. It consists of 45 items across seven subscales and two aspects of mastery motivation. Instrumental mastery focuses on persistence with tasks and includes the subscales of object-oriented persistence, gross motor persistence, social persistence with adults and social persistence with peers. Expressive mastery comprises subscales of negative reactions to failure and mastery pleasure. The final subscale, competence, is considered a separate construct which measures the child's ability to master tasks relative to peers. This involves rating each of the 45 items on a five-point scale ranging from 1=not at all typical to 5=very typical.
"change" Test of Playfulness (ToP) | Intensive and CIT Model Program: baseline, 1 week, 2 months, 6 months; Distributed CIT Model Program: baseline, 1 months, 2 months, 6 months
  The ToP is an assessment designed for measuring the playfulness of individuals between the ages 6 months and 18 years. It is composed of 24 items that are scored following an observation of the individual's free play. Items are scored on a 4-point Likert scale with respect to three dimensions: Extent (0 = rarely or never, 3 = almost always), Intensity (0 = not, 3 = highly), and Skillfulness (0 = unskilled, 3 = highly skilled).
"change" Pediatric Engagement Questionnaire (PEQ) | Intensive and CIT Model Program: baseline, 1 week, 2 months, 6 months; Distributed CIT Model Program: baseline, 1 months, 2 months, 6 months
  The PEO includes two versions, that is, child version and therapist version (PEQ-C, PEQ-T). The items of the PEQ are modified from existing questionnaires Pediatric Motivation Scale (PMOT) and based on tenets of self-determination theory. The PEQ-C consists 16 items by 5-point Likert scale with smiley face figures. It is an event-based measurement of motivation and is designed to measure motivation and the experience of receiving specific therapeutic activities. The PEQ-T represents therapists' observations of the child's engagement, participation, and persistence of master the tasks during interventions sessions. It is also designed as 5-point Likert scale on child's engagement, participation, and task persistence for therapists' points of view.
"change" Client Satisfaction Questionnaire (CSQ) | Intensive and CIT Model Program: baseline, 1 week, 2 months, 6 months; Distributed CIT Model Program: baseline, 1 months, 2 months, 6 months
  The CSQ has 24 items and 2 open-ended questions that is designed to obtain the information from the parents including their general satisfaction with service, their perspective of the intervention, their thoughts to the treatment content, dose and the importance of the intervention. The CSQ can easily be supplemented by open-ended questions and items of special interest to a particular service program, without undue time demand on clients.
"change" Parenting Stress Index-Short Form (PSI-SF) | Intensive and CIT Model Program: baseline, 1 week, 2 months, 6 months; Distributed CIT Model Program: baseline, 1 months, 2 months, 6 months
  The PSI-SF is direct derivative from the Parenting Stress Index (PSI) full-length test which was created to sample a diverse range of potential influences on parenting practices to address the need for a psychometrically sound but brief screening measure of parenting stress. All 36 items of the PSI-SF consist of three subscales: Parental Distress, Parent-Child Dysfunctional Interaction, and Difficult Child. Each subscale consists of 12 items rated from 1 (strongly disagree) to 5 (strongly agree).

CONTACTS AND LOCATIONS:
Overall Officials: Tien-Ni Wang, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Zhongzheng District, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wang TN, Liang KJ, Liu YC, Shieh JY, Chen HL. Effects of Intensive Versus Distributed Constraint-Induced Movement Therapy for Children With Unilateral Cerebral Palsy: A Quasi-Randomized Trial. Neurorehabil Neural Repair. 2023 Feb-Mar;37(2-3):109-118. doi: 10.1177/15459683231162330. Epub 2023 Mar 28. PMID 36987387